CLINICAL TRIAL: NCT03910335
Title: Diagnostic Screening Tool for Lumbar Spinal Stenosis
Acronym: LSS Screen
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: 10.180
Record Dates: First submitted 2019-04-05; First posted 2019-04-10 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LSS patients: Case/control study: Patients from surgical departments awaiting surgery for LSS will will out the questionnaire.
  Cohort study: Patients from a medical department will fill out the questionnaire, and a clinician will determine if LSS is present (reference standard)
  Interventions: Diagnostic Test: LSS Screen
- Non-LSS patients: Case/control study and cohort study: Patients from a medical department will fill out the questionnaire, and a clinician will determine if LSS is present (reference standard)
  Interventions: Diagnostic Test: LSS Screen

INTERVENTIONS:
Diagnostic Test: LSS Screen — Patients will fill out a questionnaire with 13 questions related to presence or absence of clinical symptoms of lumbar spinal stenosis (neurogenic claudication)

SUMMARY:
The aim of this project is to develop a questionnaire that should distinguish patients with lumbar spinal stenosis (LSS) from other patients. LSS can cause significant pain and disability leading to dramatically reduced quality of life, immobility and functional limitation.

The number of people with pain and disability due to LSS is expected to increase with age due to the degenerative nature of the disease. With an aging population this could potentially become a major health economic challenge.

One of the challenges to estimate the true prevalence is the lack of a valid and reliable gold standard for LSS. To our knowledge, no diagnostic screening tool designed to estimate the prevalence of LSS in a clinical population of Danish patients with chronic low back pain (LBP) and leg pain has been developed.

The objective of this project is to develop a diagnostic screening tool for LSS - the LLS Screen. This should consist of a set of items useable in a self-administered questionnaire, a rule to compute the probability of having LSS, and a cutpoint to be used to obtain a sensitivity of 95%. The rule should be applicable in patient populations suffering from low back pain and with increased suspicion to suffer from LSS due to failure of non-surgical treatment

DETAILED DESCRIPTION:
The specific objectives are:

A. To identify items with high content validity for diagnosing LLS B. To investigate the preliminary value of items included in the LLS screen C. To investigate the performance of the included items in the LLS screen D. To decide on the content of the final version of the LLS Screen

This project consists of four parts. Part I addresses objective A based on a literature search and qualitative semi-structured interviews. Part II addresses objective B by conducting a case-control study concurrent with a cohort study and performing a series of analyses to investigate the preliminary value and performance of the items. Part III describes the performance of the items by combining them in various ways to obtain an optimal diagnostic rule (objective C). Finally, part IV is a decision of the content of the final version of the LSS Screen based on information from Part I, II and III (objective D).

Part II:

A case-control study with cases and controls identified within a prospective clinical population based cohort study that will be boosted with cases of LSS.

Cohort design First, a prospective clinical population based cohort of patients with low back pain and/or leg pain will be initiated. Patients above 50 years of age will be included in the study at their first visit at the Spine Centre where they fill out the screening questionnaire (index test) before they are seen by a clinician. The primary diagnosis (reference test) will be assessed and determined by specialists at the Spine Centre.

Case-control design Secondly, patients with LSS will be recruited from other departments to artificially increase the prevalence of LSS. Patients with LSS will be recruited from the surgical department at the Spine Centre of Southern Denmark, Middelfart, Denmark and Department of Spine Surgery, Odense University Hospital (OUH), Odense, Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and write Danish
* Age above 50
* Low back pain and/or leg pain

Exclusion Criteria:

• None

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Case/control design:
  90-100 cases will be collected at surgical departments from patients assigned to surgery due to clinical symptoms of lumbar spinal stenosis
  Cohort design:
  Patients reffered from primary care to a publicly-funded outpatient secondary care spine clinic with primary compain of low back pain and/or leg pain
Sampling Method: Probability Sample
Enrollment: 383 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-10-23 (Actual)

PRIMARY OUTCOMES:
Accuracy of the screening questionnaire for lumbar spinal stenosis (LLS screen) | Baseline
  To estimate the accuracy of the questionnaire LSS Screens ability to identify patients with clinical symptoms of LSS in terms of sensitivity, specificity and diagnostic odds ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Rikke K Jensen, PhD, Principal Investigator — University of Southern Denmark (SDU)
Locations (1):
- University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Full project protocol — http://spoergeskemaer.dk/lss-screen